CLINICAL TRIAL: NCT01546701
Title: Buprenorphine in Acute Renal Colic Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 130-1848
Record Dates: First submitted 2012-03-01; First posted 2012-03-07 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Acute Pain Management; Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Renal Colic Patients treated by 2 mg sublingual Buprenorphine.
  Interventions: Drug: Buprenorphine
- Morphine (Active Comparator): Renal Colic Patients treated by 0.1 mg/kg intravenous morphine.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Buprenorphine — 2 mg sublingual tablet
  Arms: Buprenorphine
Drug: Morphine — 0.1 mg/kg IV morphine
  Arms: Morphine

SUMMARY:
The purpose of this study is to determine whether sublingual Buprenorphine is as effective as Iv Morphine sulfate on pain control of the patients with acute renal colic in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of acute renal colic; positive urinalysis of hematuria; pain score more than 3 in Numerical Rating Score (NRS); patients sign the informed consent to enroll.

Exclusion Criteria:

* previous history of seizures; cardiovascular, hepatic, renal or metabolic diseases;
* febrile patients (T > 38°C);
* hemodynamically unstable patients ( Systolic Blood Pressure < 90 mmHg);
* pregnant patients;
* patients with abdominal tenderness as a sign of peritoneal inflammation;
* any clinical suspicion for diseases other than urolithiasis like abdominal aortic aneurysm or dissection;
* patients with a history of drug addiction or known allergy to opioids;
* patients who had used analgesics 6 hours before arriving.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change in pain score | 20 and 40 minutes
  change in pain severity based on Numerical Rating Score

SECONDARY OUTCOMES:
treatment side effects | 40 minutes
  experiencing any side effects by the patients as a result of treatment protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Jalili, MD, Study Director — TUMS
Locations (1):
- TUMS, Tehran, Tehran Province, Iran